CLINICAL TRIAL: NCT00927719
Title: A Phase IV Enhanced Safety Surveillance Study of ACAM2000® in Military Personnel
Brief Title: Safety Surveillance Study of ACAM2000® Vaccinia Vaccine
Status: Completed | Type: Observational
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Other Study IDs: H-406-005
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Smallpox
Keywords: Smallpox; Smallpox Vaccine; Vaccinia virus; Military
MeSH Terms: conditions — Smallpox; Vaccinia | interventions — ACAM2000

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ACAM2000® vaccinia vaccine Cohort: Participants had received ACAM2000®, vaccinia virus Smallpox vaccine.
  Interventions: Biological: ACAM2000® smallpox vaccine

INTERVENTIONS:
Biological: ACAM2000® smallpox vaccine — Previous vaccination, no vaccine is administered in this study.
  Other Names: ACAM2000®

SUMMARY:
This is an enhanced safety surveillance study that will occur within the military Service Member population.

Primary Objective:

* To evaluate the rates of suspected, probable, and confirmed myocarditis and/or pericarditis in temporal association with ACAM2000® vaccination.

Secondary Objectives:

* To evaluate the rates of cardiovascular adverse events in temporal association with ACAM2000® vaccination.
* To evaluate the rates of neurological adverse events in temporal association with ACAM2000® vaccination.

DETAILED DESCRIPTION:
The Armed Forces Health Surveillance Activity (AFHSA) will perform comprehensive health surveillance through the operation of the Defense Medical Surveillance System (DMSS). Demographic and medical information gathered within monthly reports from the DMSS will be collected from approximately 100,000 to 200,000 military Service Members who received the ACAM2000® smallpox vaccine.

ELIGIBILITY:
Inclusion Criteria :

* Male and female military personnel >= 17 years of age.
* Have received the ACAM2000® smallpox vaccine.

Exclusion Criteria :

* Not applicable.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants that had received ACAM2000®, vaccinia virus Smallpox vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 897227 (Actual)
Dates: Start 2008-12; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the safety following vaccination with ACAM2000® vaccinia vaccine | Entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Emergent BioSolutions
Locations (4):
- United States (4):
  - Twentynine Palms, California
  - Fort Campbell North, Kentucky
  - Fort Bliss, Texas
  - Fort Hood, Texas

REFERENCES:
- [Derived] Decker MD, Garman PM, Hughes H, Yacovone MA, Collins LC, Fegley CD, Lin G, DiPietro G, Gordon DM. Enhanced safety surveillance study of ACAM2000 smallpox vaccine among US military service members. Vaccine. 2021 Sep 15;39(39):5541-5547. doi: 10.1016/j.vaccine.2021.08.041. Epub 2021 Aug 26. PMID 34454787